CLINICAL TRIAL: NCT04670107
Title: The Combination of Anlotinib and Immune Checkpoint Inhibitors for Progressed NSCLC Patients With Muti-line Therapy : a PhaseⅠB Clinical Study
Brief Title: The Combination of Anlotinib and Immune Checkpoint Inhibitors for Advanced NSCLC Patients With Muti-line Therapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, zhangxiaochun, Professor, The Affiliated Hospital of Qingdao University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANLOIM
Record Dates: First submitted 2020-11-27; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: NSCLC; Angiogenesis; Immunotherapy
MeSH Terms: interventions — anlotinib; Immune Checkpoint Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- combination group (Experimental)
  Interventions: Drug: Anlotinib in combination with Immune checkpoint inhibitors

INTERVENTIONS:
Drug: Anlotinib in combination with Immune checkpoint inhibitors — Enrolled patients received anlotinib plus Pembrolizumab treatment (anlotinib, 8-12mg, qd, 2 weeks in a row and 1 week off; anti-PD1 injection or anti-PDL1 injection, Following instructions, iv.)

SUMMARY:
Immunotherapy has made a major progress in Lung cancer.However, challenges such as primary and acquired resistance, small fraction of benefit population and lack of predictive and prognostic biomarkers even exist. The overall objective response rate is lower than 20% in second line-treatment and the progression-free survival (PFS) is also similar to or poorer than that of conventional second-line chemotherapy. Anlotinib is a novel, orally administered, multitarget receptor tyrosine kinase inhibitor that inhibits VEGFR, PDGFR, FGFR, c-Kit, and other kinases. It functions by inhibiting tumor angiogenesis and proliferative signaling pathways. We would observe and analyze the effectiveness and safety of anlotinib combined with Immune checkpoint inhibitors for advanced NSCLC after muti-line therapy to explore the synergistic effect of anti-angiogenic agents and immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form

  * Ability to comply with protocol
  * Aged ≥ 18 years Histologically documented NSCLC that is currently locally advanced or metastatic NSCLC Disease progression during or following at least one line treatment. Measurable disease, as defined by RECIST v1.1
  * ECOG performance status of 0 or 1
  * Life expectancy ≥ 12 weeks
  * Adequate hematologic and end organ function, defined by the following laboratory results obtained within 14 days prior to the first study treatment: ANC ≥ 1.5 × 109/L (without granulocyte colony-stimulating factor support within 2 weeks of laboratory test used to determine eligibility) WBC counts > 2.5 × 109/L and < 15 × 109/L Lymphocyte count ≥ 0.5 × 109/L Serum albumin ≥ 2.5 g/dL Platelet count ≥ 100 × 109/L (without transfusion within 2 weeks of laboratory test used to determine eligibility) Hemoglobin ≥ 9.0 g/dL Patients may be transfused or receive erythropoietic treatment to meet this criterion.

Liver function tests meeting one of the following criteria:

AST or ALT ≤ 2.5 × upper limit of normal (ULN), with alkaline phosphatase ≤ 2.5 × ULN or AST and ALT ≤ 1.5 × ULN in conjunction with alkaline phosphatase > 2.5 × ULN Serum bilirubin ≤ 1.5 × ULN Patients with known Gilbert's disease who have serum bilirubin level ≤ 3 × ULN may be enrolled. INR and aPTT ≤ 1.5 × ULN This applies only to patients who are not receiving therapeutic anticoagulation; patients receiving therapeutic anticoagulation should be on a stable dose for at least 1 week prior to randomization. Creatinine clearance ≥ 30 mL/min Cockcroft-Gault, Chronic Kidney Disease Epidemiology Collaboration, or Modification of Diet in Renal Disease formulas may be used for creatinine clearance calculation. Note that 24-hour urine collection is not required but is allowed.

Exclusion Criteria:

* Active or untreated CNS metastases as determined by computed tomography (CT) or magnetic resonance imaging (MRI) evaluation during screening and prior radiographic assessments Leptomeningeal disease • Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures Uncontrolled hypertension Perior used anti-angiogenic agents or immune checkpoint inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  the progression-free survival
OS | From date of randomization until the date of death from any cause, whichever came first, assessed up to 100 months
  the over survival
AE | through study completion, an average of 1 year
  adverse event caused by the combination

CONTACTS AND LOCATIONS:
Overall Officials: Zhang, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The Affiliated Hospital of Qingdao University, Qingdao, China